CLINICAL TRIAL: NCT05794191
Title: Assessment of 13-valent Pneumococcal Conjugate Vaccine Effectiveness Among People With HIV in the United States
Brief Title: A Study To Learn About The Effects Of Pneumococcal Vaccine In People With HIV
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1851217; NCT05794191 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: HIV; Pneumonia; Infections, Pneumococcal
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Persons living with HIV (PLWH): Adults with HIV
  Interventions: Biological: Vaccine Administration

INTERVENTIONS:
Biological: Vaccine Administration — PCV13 administration

SUMMARY:
The purpose of this study is to learn about how well a vaccine (Prevnar 13, PCV13) works in preventing disease in adults with HIV.

The diseases studied are pneumonia. Mostly the ones caused by the bacteria - pneumococcus. This study also evaluates the type of pneumonia that is spread into the bloodstream.

All participants in the study will be identified in health care databases. Adults with HIV will be identified by looking for a medical diagnosis that has confirmed HIV from the databases. Vaccination will be identified in the databases by looking for vaccine administration or for PCV13.

Participants will be followed in the databases to see if they have one of the diseases mentioned above or not. The number of vaccinated participants with the diseases will be compared to the number participants without the vaccines but with the diseases. This will help to understand how well the vaccine worked.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection defined as at least one inpatient or ≥2 outpatient codes related to HIV at least 30 days but no more than 730 days apart
2. At least 18 years of age at the time of the first HIV-related code
3. At least six months of continuous enrollment in medical and pharmacy plans after the first HIV-related code

Exclusion Criteria:

1. Evidence of PCV13 vaccination before the first HIV-related code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with HIV in a healthcare administrative database
Sampling Method: Non-Probability Sample
Enrollment: 350399 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1851217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data was collected from participants living with human immunodeficiency virus (PLWH) having an HIV diagnosis code between January 1, 2014 and December 31, 2021. Data was analyzed over 73 weeks in this retrospective study from March 22, 2023 to August 15, 2024.
Pre-assignment Details: A total of 350399 participants were enrolled in the study. The six months of continuous enrollment in medical and pharmacy plans between 01-Jan-2014 and 31-Dec-2021 was considered the baseline period. The end of the study occurred on the last date that administrative claims data were available on September 30, 2022. Participants were followed up from index date to the earliest of death, end of health plan enrollment or end of study period (maximum up to 8.25 years).
Groups:
- PCV13-vaccinated Participants: Participants with an HIV diagnosis code who received 13-valent pneumococcal conjugate vaccine (PCV13) were included. The participants were followed up in the databases from 14 days after their PCV13 or index date if vaccinated during the baseline period, until the earliest occurrence of outcome, death, end of health plan enrollment, or end of study period.
- Unvaccinated Participants: Participants with an HIV diagnosis code who did not receive PCV13 were included. The participants were followed in the databases from index date until the earliest occurrence of PCV13 vaccination, death, end of health plan enrollment or end of study period.
Period: Overall Study
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Started | 29435 (Number of vaccinated participants at index date, which was defined as the last day of baseline period.) | 320964 (Number of unvaccinated participants at index date, which was defined as the last day of baseline period.)
Completed | 29435 | 320964
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study. Baseline characteristics were analyzed in participants with vaccinated (PCV13 vaccinated participants) and unvaccinated (Unvaccinated participants) status at the index date, which was defined as the last day of baseline period.
Groups:
- PCV13-vaccinated Participants: Participants with an HIV diagnosis code who received PCV13 were included. The participants were followed up in the databases from 14 days after their PCV13 or index date if vaccinated during the baseline period, until the earliest occurrence of outcome, death, end of health plan enrollment, or end of study period.
- Total: Total of all reporting groups
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants | Total
Number analyzed (Participants) | 29435 | 320964 | 350399
Age, Customized [Count of Participants; unit: Participants]
  18-49 Years | 20571 | 189050 | 209621
  50-64 Years | 7907 | 113632 | 121539
  65-74 Years | 814 | 14617 | 15431
  75 Years or above | 143 | 3665 | 3808
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 22736 | 221640 | 244376
  Female | 6699 | 99319 | 106018
  Unknown | 0 | 5 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: PCV13 Vaccine Effectiveness (VE) for First Event of Invasive Pneumococcal Disease (IPD): Overall Follow-up
Description: VE:[(1-hazard ratio (HR)]*100 and was obtained from marginal structural Cox models(Cox-MSM) after applying Inverse probability of treatment (IPT)*Inverse probability of censoring(IPC)weights.IPTW was generated from predicted probabilities of vaccination status (propensity scores) to create pseudo-populations where any imbalances in potential confounders by vaccination status were reduced. IPCW was used to adjust for informative censoring. IPD: based on International Classification of Diseases,9th revision, Clinical Modification(ICD-9-CM)or ICD-10-CM.Data for total number of participants with IPD is reported in descriptive and VE (IPTW*IPCW+imbalanced variables) is reported in statistical section.PCV13 vaccination status was a time varying exposure (i.e.,vaccination status was not fixed at start of follow-up and participants could receive PCV13 during follow-up).
Time Frame: From index date to the earliest of death, end of health plan enrollment or end of study period (maximum up to 8.25 years)
Population: PCV13 vaccination status was a time varying exposure and participants could be counted in both PCV13 vaccinated or unvaccinated arms, depending on vaccination status during follow-up. Here, 'Overall Number of Participants Analyzed (N)' for Unvaccinated arm=participants unvaccinated at start of study evaluable for this outcome measure (OM); N for vaccinated arm=participants vaccinated by end of follow up for this OM; hence, N is different from those reported under participant flow and baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 85584 | 320959
Participants | 167 [57.233 to 77.529] | 747 [91.165 to 105.226]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = 22.438, 95% CI 2-sided [5.425 to 36.391]

2. Primary Outcome: VE for First Event of IPD at 0-3 Years of Follow-up
Description: VE: [(1- hazard ratio (HR)] * 100 and was obtained from Cox-MSM after applying the IPT *IPC weights. IPTW was generated from predicted probabilities of vaccination status (propensity scores) to create pseudo-populations where any imbalances in the potential confounders by vaccination status were reduced. IPCW was used to adjust for informative censoring. IPD was identified based on ICD-9-CM or ICD-10-CM codes. Data for total number of participants with episodes of IPD is reported in the descriptive section and data for vaccine effectiveness (IPTW*IPCW + imbalanced variables) is reported in statistical analysis section. PCV13 vaccination status was a time varying exposure (i.e.,vaccination status was not fixed at start of follow-up and participants could receive PCV13 during follow-up).
Time Frame: 0 to 3 years of follow up
Population: PCV13 vaccination status was a time varying exposure and participants could be counted in both PCV13 vaccinated or unvaccinated arms, depending on vaccination status during follow-up. Here, 'Overall Number of Participants Analyzed (N)' for Unvaccinated arm=participants unvaccinated at start of study evaluable for this OM; N for vaccinated arm=participants vaccinated by end of follow up for this OM; hence, N is different from those reported under participant flow and baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 75382 | 320959
Participants | 73 [47.288 to 74.868] | 566 [96.120 to 113.340]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = 34.985, 95% CI 2-sided [13.249 to 51.275]

3. Primary Outcome: VE for First Event of IPD at 3-5 Years of Follow-up
Description: Vaccine effectiveness was calculated as [(1- hazard ratio (HR)] * 100 and was obtained from Cox-MSM after applying the IPT *IPC weights. IPTW was generated from predicted probabilities of vaccination status (propensity scores) to create pseudo-populations where any imbalances in the potential confounders by vaccination status were reduced. IPCW was used to adjust for informative censoring. IPD was identified based on ICD-9-CM or ICD-10-CM codes. Data for total number of participants with episodes of IPD is reported in the descriptive section and data for vaccine effectiveness (IPTW*IPCW + imbalanced variables) is reported in statistical analysis section. PCV13 vaccination status was a time varying exposure (i.e.,vaccination status was not fixed at start of follow-up and participants could receive PCV13 during follow-up).
Time Frame: 3 to 5 years of follow up
Population: PCV13 vaccination status was a time varying exposure and participants could be counted in both PCV13 vaccinated or unvaccinated arms, depending on vaccination status during follow-up. Here, 'N' for Unvaccinated arm=number of participants unvaccinated at start of specified follow-up time evaluable for this OM; N for vaccinated arm=participants vaccinated by end of follow up time for this OM; hence, N is different from those reported under participant flow and baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 47501 | 98677
Participants | 59 [65.536 to 109.273] | 116 [69.578 to 100.157]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = -5.284, 95% CI 2-sided [-50.408 to 26.302]

4. Primary Outcome: VE for First Event of IPD at 5-7 Years of Follow-up
Description: as for outcome 3
Time Frame: 5 to 7 years of follow up
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 31770 | 48523
Participants | 32 [48.640 to 97.486] | 54 [61.365 to 104.724]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = 9.274, 95% CI 2-sided [-46.883 to 43.961]

5. Primary Outcome: PCV13 VE for First Event of Pneumococcal Pneumonia (PP): Overall Follow-up
Description: Vaccine effectiveness was calculated as [(1- hazard ratio (HR)] * 100 and was obtained from Cox-MSM after applying the IPT *IPC weights. IPTW was generated from predicted probabilities of vaccination status (propensity scores) to create pseudo-populations where any imbalances in the potential confounders by vaccination status were reduced. IPCW was used to adjust for informative censoring. PP was identified based on ICD-9-CM or ICD-10-CM codes. Data for total number of participants with episodes of PP is reported in the descriptive section and data for vaccine effectiveness (IPTW*IPCW + imbalanced variables) is reported in statistical analysis section. PCV13 vaccination status was a time varying exposure (i.e.,vaccination status was not fixed at start of follow-up and participants could receive PCV13 during follow-up).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 85487 | 320959
Participants | 309 [110.734 to 138.408] | 1362 [169.723 to 188.744]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = 17.169, 95% CI 2-sided [3.994 to 28.536]

6. Primary Outcome: VE for First Event of PP at 0-3 Years of Follow-up
Description: Vaccine effectiveness was calculated as [(1- hazard ratio (HR)] * 100 and was obtained from Cox-MSM after applying the IPT *IPC weights. IPTW was generated from predicted probabilities of vaccination status (propensity scores) to create pseudo-populations where any imbalances in the potential confounders by vaccination status were reduced. IPCW was used to adjust for informative censoring. PP was identified based on ICD-9-CM or ICD-10-CM codes. Data for total number of participants with episodes of PP is reported in the descriptive section data for vaccine effectiveness (IPTW*IPCW + imbalanced variables) is reported in statistical analysis section. PCV13 vaccination status was a time varying exposure (i.e.,vaccination status was not fixed at start of follow-up and participants could receive PCV13 during follow-up).
Time Frame: 0 to 3 years of follow up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 75322 | 320959
Participants | 161 [113.143 to 154.129] | 1092 [190.119 to 214.066]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = 25.526, 95% CI 2-sided [9.400 to 38.781]

7. Primary Outcome: VE for First Event of PP at 3-5 Years of Follow-up
Description: as for outcome 5
Time Frame: 3 to 5 years of follow up
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 47365 | 98430
Participants | 94 [110.920 to 166.264] | 184 [115.149 to 153.758]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = -7.561, 95% CI 2-sided [-42.076 to 18.569]

8. Primary Outcome: VE for First Event of PP at 5-7 Years of Follow-up
Description: as for outcome 5
Time Frame: 5 to 7 years of follow up
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 31660 | 48369
Participants | 49 [80.542 to 141.172] | 69 [81.402 to 130.586]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = 11.442, 95% CI 2-sided [-34.916 to 41.871]

9. Primary Outcome: PCV13 VE for First Event of All-cause Pneumonia (ACP): Overall Follow-up
Description: Vaccine effectiveness was calculated as [(1- hazard ratio (HR)] * 100 and was obtained from Cox-MSM after applying the IPT *IPC weights. IPTW was generated from predicted probabilities of vaccination status (propensity scores) to create pseudo-populations where any imbalances in the potential confounders by vaccination status were reduced. IPCW was used to adjust for informative censoring. ACP was identified based on ICD-9-CM or ICD-10-CM codes. Data for total number of participants with episodes of ACP is reported in the descriptive section and data for vaccine effectiveness (IPTW*IPCW + imbalanced variables) is reported in statistical analysis section. PCV13 vaccination status was a time varying exposure (i.e.,vaccination status was not fixed at start of follow-up and participants could receive PCV13 during follow-up).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 80591 | 320959
Participants | 8098 [3637.505 to 3799.459] | 34498 [4922.665 to 5027.661]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = 8.435, 95% CI 2-sided [5.705 to 11.086]

10. Primary Outcome: VE for First Event of ACP at 0-3 Years of Follow-up
Description: as for outcome 9
Time Frame: 0 to 3 years of follow up
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 72303 | 320959
Participants | 4543 [3903.147 to 4136.881] | 27984 [5433.501 to 5562.327]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = 11.445, 95% CI 2-sided [8.089 to 14.679]

11. Primary Outcome: VE for First Event of ACP at 3-5 Years of Follow-up
Description: as for outcome 9
Time Frame: 3 to 5 years of follow up
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 41296 | 86841
Participants | 2079 [3405.879 to 3711.656] | 4437 [3636.291 to 3856.707]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = 7.125, 95% CI 2-sided [1.427 to 12.493]

12. Primary Outcome: VE for First Event of ACP at 5-7 Years of Follow-up
Description: Vaccine effectiveness was calculated as [(1- hazard ratio (HR)] * 100 and was obtained from Cox-MSM after applying the IPT *IPC weights. IPTW was generated from predicted probabilities of vaccination status (propensity scores) to create pseudo-populations where any imbalances in the potential confounders by vaccination status were reduced. IPCW was used to adjust for informative censoring. ACP was identified based on ICD-9-CM or ICD-10-CM codes. Data for total number of participants with episodes of ACP is reported in the descriptive section and data for vaccine effectiveness (IPTW*IPCW + imbalanced variables) is reported in statistical analysis section. PCV13 vaccination status was a time varying exposure (i.e.,vaccination status was not fixed at start of follow-up and participants could receive PCV13 during follow-up.
Time Frame: 5 to 7 years of follow up
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 25890 | 40301
Participants | 1200 [3132.249 to 3507.557] | 1757 [3101.962 to 3406.066]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; Test type: Superiority; Vaccine effectiveness percentage = -3.716, 95% CI 2-sided [-12.626 to 4.488]

13. Secondary Outcome: PCV13 VE for First Event of Pneumococcal Pneumonia or Pneumonia With Unspecified Causes at 0-3, 3-5, 5-7 and Overall Years of Follow-up
Description: Vaccine effectiveness was calculated as [(1- hazard ratio (HR)] * 100 and was obtained from Cox-MSM after applying the IPT *IPC weights. IPTW was generated from predicted probabilities of vaccination status (propensity scores) to create pseudo-populations where any imbalances in the potential confounders by vaccination status were reduced. IPCW was used to adjust for informative censoring. Data for total number of participants with episodes of pneumococcal pneumonia or pneumonia with unspecified causes are reported in the descriptive section and data for vaccine effectiveness (IPTW*IPCW + imbalanced variables) is reported in statistical analysis section. PCV13 vaccination status was a time varying exposure (i.e.,vaccination status was not fixed at start of follow-up and participants could receive PCV13 during follow-up).
Time Frame: 0 to 3 years, 3 to 5 years and 5 to 7 years of follow-up (maximum up to 8.25 years)
Population: PCV13 vaccination status was a time varying exposure and participants could be counted in both PCV13 vaccinated or unvaccinated arms, depending on vaccination status during follow-up. Here, 'N' for Unvaccinated arm=participants unvaccinated at start of study evaluable for this OM; N for vaccinated arm=participants vaccinated by end of follow up for this OM; hence, N is different from those reported under participant flow and baseline. ."n":number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 81338 | 320959
Participants
  0-3 Years: number analyzed (Participants) | 72833 | 320959
  0-3 Years | 3996 [3384.055 to 3600.551] | 24423 [4694.780 to 4814.028]
  3-5 Years: number analyzed (Participants) | 42096 | 88266
  3-5 Years | 1886 [3016.434 to 3301.388] | 3979 [3193.903 to 3398.684]
  5-7 Years: number analyzed (Participants) | 26564 | 41224
  5-7 Years | 1031 [2597.852 to 2935.209] | 1460 [2496.416 to 2766.140]
  Overall follow up | 7155 [3147.928 to 3297.244] | 30139 [4242.686 to 4339.574]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; IPTW*IPCW + imbalanced variables: 0-3 years; Test type: Superiority; Vaccine effectiveness percentage = 13.685, 95% CI 2-sided [10.213 to 17.022]
Statistical Analysis 2: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; IPTW*IPCW + imbalanced variables: 3-5 years; Test type: Superiority; Vaccine effectiveness percentage = 7.665, 95% CI 2-sided [1.707 to 13.261]
Statistical Analysis 3: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; IPTW*IPCW + imbalanced variables: 5-7 years; Test type: Superiority; Vaccine effectiveness percentage = -5.792, 95% CI 2-sided [-15.691 to 3.260]
Statistical Analysis 4: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; IPTW*IPCW + imbalanced variables: overall follow up; Test type: Superiority; Vaccine effectiveness percentage = 9.902, 95% CI 2-sided [7.056 to 12.660]

14. Secondary Outcome: PCV13 VE for First Event of Pneumonia With Unspecified Causes at 0-3, 3-5, 5-7 and Overall Years of Follow-up
Description: VE was calculated as [(1-hazard ratio (HR)] * 100 and was obtained from Cox-MSM after applying the IPT *IPC weights. IPTW was generated from predicted probabilities of vaccination status (propensity scores) to create pseudo-populations where any imbalances in the potential confounders by vaccination status were reduced. IPCW was used to adjust for informative censoring. Pneumonia with unspecified causes was identified based on ICD-9-CM or ICD-10-CM codes. Data for total number of participants with episodes of pneumonia with unspecified causes are reported in the descriptive section and data for vaccine effectiveness (IPTW*IPCW + imbalanced variables) is reported in statistical analysis section. PCV13 vaccination status was a time varying exposure (i.e.,vaccination status was not fixed at start of follow-up and participants could receive PCV13 during follow-up).
Time Frame: 0 to 3 years, 3 to 5 years and 5 to 7 years of follow-up (maximum up to 8.25 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
Number analyzed (Participants) | 81361 | 320959
Participants
  0-3 Years: number analyzed (Participants) | 72853 | 320959
  0-3 Years | 3980 [3368.927 to 3584.902] | 24302 [4669.755 to 4788.667]
  3-5 Years: number analyzed (Participants) | 42120 | 88312
  3-5 Years | 1881 [3006.512 to 3290.923] | 3970 [3184.563 to 3388.983]
  5-7 Years: number analyzed (Participants) | 26581 | 41255
  5-7 Years | 1030 [2593.321 to 2930.264] | 1461 [2496.054 to 2765.642]
  Overall follow up | 7133 [3136.465 to 3285.472] | 30010 [4222.550 to 4319.187]
Statistical Analysis 1: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; IPTW*IPCW + imbalanced variables: 0-3 years; Test type: Superiority; Vaccine effectiveness percentage = 13.631, 95% CI 2-sided [10.149 to 16.978]
Statistical Analysis 2: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; IPTW*IPCW + imbalanced variables: 3-5 years; Test type: Superiority; Vaccine effectiveness percentage = 7.673, 95% CI 2-sided [1.708 to 13.276]
Statistical Analysis 3: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; IPTW*IPCW + imbalanced variables: 5-7 years; Test type: Superiority; Vaccine effectiveness percentage = -5.897, 95% CI 2-sided [-15.809 to 3.166]
Statistical Analysis 4: Comparison: PCV13-vaccinated Participants vs Unvaccinated Participants; IPTW*IPCW + imbalanced variables: overall follow up; Test type: Superiority; Vaccine effectiveness percentage = 9.853, 95% CI 2-sided [7.000 to 12.617]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events were not planned to be collected; hence, time frame was not applicable.
Description: In this observational retrospective study of deidentified database individual identifying information was not available. Minimum criteria for reporting an adverse event could not be met, hence all-cause mortality, serious adverse events (SAEs) and other AEs were not planned to be collected. Thus reporting "0" participants at risk.
Arm/Group | PCV13-vaccinated Participants | Unvaccinated Participants
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT05794191/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT05794191/SAP_001.pdf